CLINICAL TRIAL: NCT06911619
Title: Impact of Nutritional Management on the Frailty of Patients Waiting for Liver Transplantation (Via the LFI Tool)
Acronym: LFI-PATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL24_1201
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Fragility; Cirrhosis; Hepatic Transplantation; Undernutrition
Keywords: nutrition; Hepatic Transplantation; Cirrhosis
MeSH Terms: conditions — Fibrosis; Malnutrition | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Prospective interventional, single-center, randomized, longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary intervention Group (Experimental): The intervention consists of a personalized dietary management with a nutritional follow-up pending transplantation. Teleconsultation appointments are scheduled with the dietician for dietary coaching and a re-evaluation of the nutritional strategy. Follow-up visits in person, carried out by the dietician at the 3rd and 6th month waiting for liver transplantation and are coupled with the usual consultations with the referring hepatologist. The visits allow the realization of LFI (Liver Frailty Index), the collection of interrelated events and the reassessment of hepatic disease as well as the re-evaluation of the nutritional strategy (oral nutritional supplement, enteral or parenteral nutrition)
  Interventions: Dietary Supplement: Dietary management
- Standard Follow up (Other): The patient will be followed up by his referee hepatologist every 3 months. The 3-month and 6-month follow-up visits pending transplantation will be performed with a Clinical Research Assistant on the same day as the follow-up consultation with his hepatologist with the completion of the LFI test and the collection of intercurrent events and the re-evaluation of the liver disease.
  Interventions: Other: No dietary management

INTERVENTIONS:
Dietary Supplement: Dietary management — The intervention consists of a personalized dietary management with a nutritional follow-up pending transplantation. Teleconsultation appointments are scheduled with the dietician for dietary coaching and a re-evaluation of the nutritional strategy every month. Follow-up visits in person, carried out by the dietitian at the 3rd and 6th month waiting for transplant and are coupled with the usual consultations with the referring hepatologist. The visits allow the realization of LFI (Liver Frailty Index), the collection of interrelated events and the reassessment of hepatic disease as well as the re-evaluation of the nutritional strategy (CNO, enteral or parenteral nutrition)
  Arms: Dietary intervention Group
Other: No dietary management — The patient will be followed up by his reference hepatologist every 3 months. Follow-up visits at 3 months and 6 months waiting for liver transplantation will be performed by Clinical Research assistant on the same day as the follow-up consultation with his hepatologist with the completion of the Liver Frailty Index test and the collection of intercurrent events and the reassessment of liver disease.
  Other Names: Liver Frailty Index
  Arms: Standard Follow up

SUMMARY:
Cirrhosis is a major public health issue responsible for about 15000 deaths each year. Liver transplantation (LT) remains the only curative treatment for decompensated cirrhosis. Decompensated cirrhotic patients awaiting LT are malnourished, sarcopenic and fragile. The evaluation of the nutritional status of these patients is complex because the anthropometric data that define undernutrition (weight variation, BMI) are often compromised by the presence of edema and ascites related to liver disease. It therefore seems appropriate to focus on the fragility and sarcopenia of the cirrhotic patient as a reflection of the nutritional status. In 2017, the American team of Lai et al. validated a Liver fraily index (LFI) score of frailty specific to cirrhotic patients waiting for LT. The LFI is composed of three simple physical tests (Grip test, chair lift test, and balance tests) performed at the patient's bedside, which results in a quantitative and reproducible frailty score. Frailty while waiting for LT is associated with an increase in mortality on the waiting list, independently of the MELD (Model for End stage Liver disease) score, which is a reflection of liver severity. About half of the patients who are candidates for LT will present an aggravation of their frailty while waiting for LT. To date, no study has reported the results of a nutritional intervention on the evolution of fragility in patients awaiting LT. The objective of our study is to evaluate the impact of a nutritional management and follow-up by a dietitian specialized in hepatology on the fragility of patients waiting for LT. This is a monocentric study, randomized in two parallel groups (an intervention group with nutritional follow-ups by a trained dietitian and a control group with follow-up by the reference hepatologist without specific dietary management by a dietician) in open. All patients enrolled on the LT list with an LFI > 3.2 (pre-frail and frail state) will be included in the study. It is planned to include 210 patients over a period of 24 months. The LFI will be measured for all patients (control group + intervention group) at 3 and 6 months, as part of their follow-up in the LT center. This study will also make it possible to correlate frailty with other parameters (severity of liver disease, access to LT).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient registered on the waiting list for Hepatic Transplantation in the Transplantation center of the Croix Rousse Hospital (GHN), Hospices Civils de Lyon
* Dated and signed an informed consent
* Affiliated to a social security scheme or beneficiary of a similar scheme

Exclusion Criteria:

* Patient hospitalized in intensive care
* Patient with initial LFI test result < to 3.2, that is considered as "robust".
* Patient unable to perform LFI exercises (chronic or acute motor disability in lower or upper limbs)
* Pregnant, parturient or lactating women
* Persons deprived of liberty by a judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Inability to understand protocol information
* Subject participating in another interventional research including an ongoing exclusion period at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact at 3 months, of a nutritional management and follow-up by a dietitian specialized in hepatology compared to the usual management without dietary follow-up, on the fragility of patients waiting for liver transplantation (LT). | 3rd month after visit 1.
  Measurement of LFI (Liver fraily index) score score variation between D0 (baseline = visit 1) and 3 months (first reassessment = visit 2) during the liver transplantation waiting period. This variation will be compared between the intervention group and the control group.

SECONDARY OUTCOMES:
Evaluate the impact of a nutritional follow-up on the fragility of patients at 6 months on list | 6th Month after visit 1.
  For patients still on the liver transplantation waiting list, comparison between the intervention and control group of the LFI (Liver fraily index) variation between Baseline (visit 1) and month 6 (visit 3).
Evaluate the impact of a nutritional follow-up on the distribution of patients' frailty according to classes: robust, pre-fragile, fragile | 3rd Month (M3) after Visit 1 and M6 after V1
  Compare the evolution of the fragility profile (Robust - Prefragile - Fragile) of patients waiting for liver transplantation according to LFI (Liver fraily index) at M3 and M6 in the intervention group and in the control, group compared with the initial LFI (D0)
Evaluate compliance with oral nutritional supplement treatment for patients awaiting transplant | 3rd Month and 6th month after Visit 1
  At each follow-up visit (M3 and M6) assessment of compliance with oral nutritional supplements for patients who were prescribed oral nutritional supplements, through questioning their intake: 0, 1⁄4, 1⁄2, 3⁄4 or all of the oral nutritional supplements consumed compared to the prescription.
Evaluate the relationship between fragility and severity of liver disease (MELD score) | Day 0, 3rd Month (M3) and 6th Month (M6)
  Measure the correlation between LFI (Liver fraily index) at Day 0, M3 and M6 and the severity of liver disease (MELD score),
Evaluate the relationship between fragility and access to a transplant | Day 0, Month 3 after Visit 1, Month 6 after Visit 1
  Measure the correlation between the LFI (Liver fraily index) score at Day 0, Month 3 and Month 6 and access to the transplant
Evaluate the relationship between fragility and mortality on waiting list of transplantation or leaving the list due to worsening | Day 0, 3rd month and 6th month
  Measure the correlation between LFI (Liver fraily index) score at Day0, M3 and M6 and on-list mortality or leaving the list due to worsening
Evaluate the relationship between frailty and unscheduled hospitalizations while waiting for Liver Transplantation | Day 0, 3rd month and 6th month after Visit 1
  Measure the correlation with the LFI (Liver fraily index) score on Day 0, M3 and M6 and unscheduled hospitalizations awaiting transplant: numbers and indications (infections, encephalopathy, hemorrhage, etc.)
Evaluate the satisfaction of dieticians in carrying out nutritional monitoring for patients waiting for liver transplantation (logistics of organizing consultations and teleconsultations) | study completion at Month 30
  Evaluate the satisfaction of dieticians in carrying out nutritional monitoring for patients waiting for Liver Transplantation (logistics of organizing consultations and teleconsultations) via questionnary

CONTACTS AND LOCATIONS:
Overall Officials: Maxime PATUREL, Principal Investigator — Service Rééducation Nutritionnelle Hôpital de la Croix Rousse / GHN
Locations (1):
- Hôpital de la Croix Rousse / GHN, Lyon, France